CLINICAL TRIAL: NCT02865577
Title: Right Heart Dysfunction and Pulmonary Hypertension Evaluation in Airway Disease Using Cardiac Magnetic Resonance
Acronym: RiPAIR
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0519; 171377 (Other: Integrated Research Application System)
Record Dates: First submitted 2016-08-02; First posted 2016-08-12 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Asthma; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Storage of plasma extracted from the blood for biomarker (characteristic biological properties or molecules detected in blood that indicate normal or diseased processes in the body) analysis at a future date to complement similar ethically approved research at University of Leicester / University Hospitals of Leicester or other United Kingdom or international academic partners. The plasma will be stored anonymously at -80°C indefinitely atthe Leicester Respiratory Biomedical Research Unit.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Adult asthma: Adult asthma subjects with airflow limitation (FEV1% predicted < 80%) will be recruited for this study.
  Participants will undergo following study assessments:
  1. Clinical History
  2. Health status and disease control questionnaires
  3. Focused physical examination
  4. Electrocardiogram (ECG)
  5. Blood test
  6. Spirometry
  7. Echocardiogram
  8. Cardiac magnetic resonance (CMR) imaging
  9. CMR survey
- Adult COPD: Adult COPD subjects with airflow limitation (FEV1% predicted < 80%) will be recruited for this study.
  Participants will undergo following study assessments:
  1. Clinical History
  2. Health status and disease control questionnaires
  3. Focused physical examination
  4. Electrocardiogram (ECG)
  5. Blood test
  6. Spirometry
  7. Echocardiogram
  8. Cardiac magnetic resonance (CMR) imaging
  9. CMR survey
- Healthy participants: Healthy participants with no past history of cardiovascular or respiratory disease.
  Participants will undergo following study assessments:
  1. Clinical History
  2. Focused physical examination
  3. Electrocardiogram (ECG)
  4. Blood test
  5. Spirometry
  6. Echocardiogram
  7. Cardiac magnetic resonance (CMR) imaging
  8. CMR survey

SUMMARY:
Poor function of the right side of the heart and rise in pressure of the blood vessels leading to the lungs are two main heart-related factors that are associated with worsening of airway disease. A relatively new method which uses magnetic field to create images of the heart called cardiac magnetic resonance (CMR) imaging shows immense promise in detailed and accurate assessment of the heart in patients with airway diseases. This project aims to assess the heart in patients with asthma and chronic obstructive pulmonary disease (COPD) as well as healthy participants using CMR to help us determine features on CMR that are different is patients with asthma and COPD compared to healthy participants. This may help with early identification of patients who are at risk of episodes of acute worsening of airway disease, called exacerbation, and potentially halt the progression of the heart dysfunction with currently available or new treatments.

Study involves one visit at Glenfiled Hospital, Leicester, lasting approximately 4 hours. The visit will include following assessments: clinical history, health status, physical examination, electrocardiogram (ECG), blood tests, lung function testing, echocardiogram and CMR. Part of the study will involve a participant questionnaire in which the participants will rate their CMR experience. The results will potentially change the way CMR is undertaken. A sub-set of the participants will also be invited back to do a one off focus group discussing the CMR experience further.

DETAILED DESCRIPTION:
Background and Importance:

Chronic respiratory diseases, which include asthma, COPD and pulmonary hypertension (PH), were responsible for 4.2 million deaths globally in 2008. COPD and asthma affect more than 500 million people worldwide and present an enormous health and economic burden.

Exacerbations of airway disease contribute to disease progression and represent a substantial proportion of acute hospital admissions. Early identification of patients at risk of such events is therefore important. There is unclear distinction between the two airway diseases, particularly in their severe form with evidence of heterogeneity. Right ventricular dysfunction(RVD) and PH secondary to lung disease and/or hypoxia are now recognised as important elements of chronic airway disease pathogenesis and play an important role in the development of frequent comorbidities. There are now data suggesting that pulmonary artery dilatation in COPD patients is associated with increased risk of exacerbations. This indicates that cardiovascular factors in addition to airway inflammation may be associated with exacerbations in airway diseases. Development of RVD and PH in COPD patients are also associated with poor exercise tolerance.RVD can be seen before the development of PH and cor pulmonale in COPD. This underpins the importance of early diagnosis as this may improve overall survival and quality of life.

Clinical diagnosis of PH in chronic airway diseases is often difficult, particularly in the mild form due to similarity in clinical presentation. Other methods for diagnosis of RVD and PH are echocardiography and right heart catheterisation(RHC). The echocardiographic measurements have been shown to lack sensitivity and specificity on patients with COPD and the RHC is an invasive test, with risk of complications. Cardiac magnetic resonance (CMR) imaging provides an excellent alternative for diagnosis of RVD and PH. CMR is a non-invasive test, free from ionizing radiation and the CMR morphometric indices have dramatically lower inter-observer and intra-observer variability and test-retest reproducibility compared to echocardiography. There is a paucity of information on the value of CMR in Group 3 PH. It is also unclear whether PH plays a role in severe asthma patients who have airway inflammation and airflow limitation comparable to COPD patients.

Study Participants:

The investigators plan to recruit a total of 86 participants for this study. Adult asthma and COPD subjects with airflow limitation (FEV1% predicted < 80%) will be recruited for this study. Healthy participants with no past history of cardiovascular or respiratory disease will also be recruited. The investigators plan to recruit 33 participants (n=13 with FEV1% predicted < 50%, n=20 with FEV1% predicted ≥ 50% and < 80%) in each group with airway disease (COPD and asthma) and 20 healthy participants.

Study Assessments:

Participants will undergo the following assessments on the day of their visit:

1. Clinical History Clinical history will be recorded as done routinely in clinics, which will include date of birth, gender, disease duration, age of onset, other medical conditions, smoking history, occupational history, severe exacerbations in last one year (requiring use of steroid tablets or emergency hospital visit) and treatment.
2. Health status and disease control questionnaires (Only for Airway Disease Participants) Participants will be asked to complete routine health status and disease control questionnaires.
3. Focused physical examination Participant's height and weight will be measured. Pulse oximetry will also be performed. Pulse oximetry is a non-invasive method to measure the oxygen level in the blood by placing a sensor device on a person's body, usually fingertip or earlobe.
4. Electrocardiogram (ECG) An ECG will be performed on all participants.
5. Blood test Blood will be obtained for the following: (1) assessment of a protein secreted by the heart chambers in response to excessive stretching of the heart muscles, (2) full blood count [FBC] (3) urea and electrolytes [U&E] and (4) storage of plasma extracted from the blood for biomarker (characteristic biological properties or molecules detected in blood that indicate normal or diseased processes in the body) analysis at a future date to complement similar ethically approved research at University of Leicester / University Hospitals of Leicester or other United Kingdom or international academic partners. The plasma will be stored anonymously at -80°C indefinitely at the NIHR Leicester Respiratory Biomedical Research Unit.
6. Spirometry Lung function of all the participants will be assessed using spirometry (breathing test).
7. Echocardiogram A focussed test will be performed to measure the pressure with the pulmonary artery
8. Cardiac magnetic resonance (CMR) imaging

   After identification of the position of the heart using localisers the following sequences will be obtained:

   (i) Cine Imaging: Biventricular volume, function and mass. Interventricular septum and left ventricle eccentricity index will be calculated. Pulmonary artery(PA) stiffness and pulsatility will be assessed by measuring the relative area change of the pulmonary trunk during the cardiac cycle.

   (ii) Phase-contrast magnetic resonance imaging(MRI) Cardiac output and flow profile will be determined. (iii) Magnetic Resonance Angiography(MRA) Contrast-enhanced MRA will be acquired to assess the pulmonary vascular tree to accurately quantify dimensions and assess angiogram pattern of the pulmonary vascular tree.

   (iv) Late Gadolinium Enhancement(LGE) T1-weighted inversion recovery gradient echo images will be acquired approximately 15-20 minutes after intravenous injection of gadolinium based contrast agent. Degree of LGE at the insertion points of the interventricular septum will be assessed.

   (v) Myocardial T1 mapping T1-mapping sequence based on Modified Look-Locker Inversion-recovery(MOLLI) technique will be used for assessment of myocardial fibrosis.
9. CMR survey A questionnaire will be given to the participants after the CMR scan to find out about their experience during the examination.

ELIGIBILITY:
Inclusion Criteria:

Airway Disease (Asthma and COPD)

1. Participant is willing and able to give informed consent for participation in the study.
2. Male or Female, aged 18 years or above.
3. Participants diagnosed with Asthma or COPD with airflow limitation (FEV1% predicted < 80%) with no exacerbations for at least 4 weeks prior to study entry.
4. Participant has no clinical contraindication for CMR scan.
5. Able (in the Investigators opinion) and willing to comply with all study requirements.
6. Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Healthy Volunteers

1. Participant is willing and able to give informed consent for participation in the study.
2. Male or Female, aged 18 years or above.
3. Healthy participant in good health with no past history of cardiovascular or respiratory disease.
4. Participant has no clinical contraindication for CMR scan.
5. Able (in the Investigators opinion) and willing to comply with all study requirements.
6. Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

Airway Disease (Asthma and COPD)

The participant may not enter the study if ANY of the following apply:

1. Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
2. Severe renal impairment eGFR < 30 ml/min.
3. Contraindication for undergoing CMR scan including permanent pacemaker and surgical procedure within last 6 weeks.
4. Unable to understand / read English
5. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Healthy Volunteers

The participant may not enter the study if ANY of the following apply:

1. Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
2. Severe renal impairment eGFR < 30 ml/min.
3. Contraindication for undergoing CMR scan including permanent pacemaker and surgical procedure within last 6 weeks.
4. Unable to understand / read English
5. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators plan to recruit a total of 86 participants for this study. Adult asthma and chronicobstructive airway disease (COPD) patients with airflow limitation (FEV1% predicted < 80%) will be recruited for this study. Healthy participants with no past history of cardiovascular or respiratory disease will also be recruited. The investigators plan to recruit 33 participants (n=13 with FEV1% predicted < 50%, n=20 with FEV1% predicted ≥ 50% and < 80%) in each group with airway disease (COPD and asthma) and 20 healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-07-02 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Right ventricle End Diastolic volume assessed by cardiac magnetic resonance | On the day of Cardiac Magnetic Resonance

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Gupta, PhD, FRCR, Principal Investigator — University of Leicester / University Hospitals of Leicester NHS Trust
Locations (1):
- Glenfield Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No